CLINICAL TRIAL: NCT05619497
Title: Offering Women PrEP With Education and Shared Decision-making (Aim 2)
Brief Title: The OPENS Trial: Offering Women PrEP (Aim 2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Florida Department of Health (Other Government); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: IRB # 2020-014-FDOH; 3R01MD013565 (NIH)
Record Dates: First submitted 2022-11-03; First posted 2022-11-17 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Human Immunodeficiency Virus; Human Immunodeficiency Virus Transmission; Sexually Transmitted Diseases
Keywords: Pre-exposure prophylaxis (PrEP); HIV prevention behaviors; HIV prevention methods; HIV education; African American, Latina, women of color; Shared decision making; Shared decision-making; Decision making, shared; Trauma informed care; Trauma-informed care; Patient decision support; Patient decision aid; Public health clinic; Health department clinic; Southeastern U.S.
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Care Post Clinic-Wide Trainings (Active Comparator): Participants in this arm will receive care in a clinic where providers and staff have been trained in shared decision making and trauma-informed care. Participants in this arm will not view the decision support tool in this phase.
  Interventions: Other: Clinic-wide Trainings
- Care Post Clinic-Wide Training and HIV Prevention Decision Support Tool (DST) (Experimental): Participants in this arm will receive care in a clinic where providers and staff have been trained in shared decision making and trauma informed care, and receive the HIV prevention DST intervention immediately before their provider visit.
  Interventions: Other: Clinic-wide Trainings and HIV Prevention Decision Support Tool (DST)
- Standard Care without the HIV Prevention Decision Support Tool (DST) (No Intervention): Participants in this arm will receive usual care at a clinic that has not received training in shared decision making and trauma-informed care. These participants also will not have viewed the HIV prevention DST. These participants were recruited in Aim 1 of this study.
- Standard care with the HIV Prevention Decision Support Tool (DST) (Active Comparator): Participants in this arm will receive usual care at a clinic that has not received training in shared decision making and trauma-informed care. These participants will view the HIV prevention DST. These participants were recruited in Aim 1 of this study.
  Interventions: Other: Standard Care with the HIV Prevention Decision Support Tool (DST)

INTERVENTIONS:
Other: Clinic-wide Trainings — The clinic-wide trainings combine principles of shared decision-making and trauma informed care to inform providers and clinic staff of an equitable approach to offering HIV prevention information. These care delivery approaches have been used in health education and counseling in a range of contexts and are effective strategies for care provision. Participants in this arm will receive care from providers and staff who received training.
  Arms: Care Post Clinic-Wide Trainings
Other: Clinic-wide Trainings and HIV Prevention Decision Support Tool (DST) — The clinic-wide trainings combine principles of shared decision-making and trauma informed care to inform providers and clinic staff of an equitable approach to offering HIV prevention information. These care delivery approaches have been used in health education and counseling in a range of contexts and are effective strategies for care provision. Participants in this arm will receive care from providers and staff who received training.
  The DST is founded on principles of decision-science and will address barriers to PrEP delivery. The DST will present HIV prevention information through a tablet in the clinical setting. The tool provides information about vulnerabilities to HIV and core characteristics of different HIV prevention methods, and the opportunity to explore these characteristics in depth, including efficacy, safety and side effects. The tool emphasizes the highly variable and individual nature of baseline risk.
  Arms: Care Post Clinic-Wide Training and HIV Prevention Decision Support Tool (DST)
Other: Standard Care with the HIV Prevention Decision Support Tool (DST) — Participants in this arm will receive usual care at a clinic that has not received training in shared decision making and trauma informed care. These participants will view the decision support tool. These participants were recruited in Aim 1 of this study.
  Arms: Standard care with the HIV Prevention Decision Support Tool (DST)

SUMMARY:
To address the significant barriers to pre-exposure prophylaxis (PrEP) implementation for cisgender women and address racial inequities in HIV prevention in the United States (US), a novel approach that accounts for multilevel influences is necessary. This study is the second part (Aim 2) of a multi-component project and involves a patient- and clinic-level intervention in a public health family planning clinic in Duval County Florida, where most patients are women of color. The area has one of the highest HIV incidence rates among women in the US. The investigators developed 1) a tablet-based decision support tool (DST) that helps users learn about HIV vulnerabilities and HIV prevention strategies to inform how they consider options for reducing their likelihood of acquiring HIV, and 2) clinic-wide trainings regarding shared decision making and trauma informed care. In Aim 1 (previously completed), participants were randomized to viewing an HIV prevention DST in a clinic that had not received clinic-wide trainings. In Aim 2 (the present study), there will be two phases. In the first phase, participants will receive care at the clinic following training; the DST will not be used. In the second phase, in addition to being seen at a clinic-site that has experienced the training, participants will use the DST before their visit. Participants will be surveyed about experiences with HIV prevention counseling, intentions about using HIV prevention, and DST use (among those in the active arm in the second phase). A subset of participants, individuals who self-identify as Black or Latinx, will also complete a post-clinic visit interview. The investigators will assess whether participants initiated an HIV prevention method three months following their initial visit. The main outcomes will include a quantitative and qualitative assessment of PrEP or other HIV prevention use, decisional certainty, and satisfaction with information about HIV prevention options.

DETAILED DESCRIPTION:
Although 13% of the U.S. female population is Black, 60% of new HIV diagnoses in U.S. women occur among Black women. The South is the epicenter of the U.S. HIV epidemic, including in women, and Black Southern women are disproportionately affected: Black women account for 69% of new HIV diagnoses in women in the South. As the first highly effective, discrete, woman-controlled HIV prevention method, oral pre-exposure prophylaxis (PrEP) with tenofovir disoproxil fumarate/emtricitabine radically expands HIV prevention options for women. However, uptake of PrEP in U.S. women has lagged, particularly among groups most affected by HIV.

PrEP cascades outline the necessary steps for accessing PrEP, including screening and identifying eligible individuals, linkage to care, prescription, and initiation of PrEP. Data suggest there are multilevel barriers related to the process of screening for HIV risk in women and identifying potential PrEP candidates that may drive a significant drop off early in the PrEP cascade for women. Women report feeling judged by risk assessment questions and experience stigma around disclosing sexual practices. As a result, if screening is required to educate patients about PrEP - as is true in most clinical settings - many women for whom PrEP is appropriate may never learn about PrEP. Further, women have low levels of knowledge about HIV risk and HIV prevention options, and therefore will not seek out PrEP services themselves. Lastly, there is often limited time to educate patients in busy clinics. By offering education to all women about vulnerabilities to HIV as well as information about HIV prevention methods including PrEP, at-risk women can circumvent these multifactorial barriers and request PrEP. Electronic decision support tools (DST), which have been used with success in a range of healthcare contexts including contraception, provide an efficient and private mechanism for this information-sharing step.

The study team developed a tablet-based tool that is designed to provide universal PrEP education and facilitate women's agency to identify their own risks and interest in PrEP. It was refined with iterative feedback from patient and community stakeholders and finalized based on cognitive testing.

The DST provides information about vulnerabilities to HIV, and emphasizes the variable and individual nature of baseline risk. It provides information on the core characteristics of different HIV prevention methods, and then the opportunity to explore these characteristics in depth, including efficacy, safety and side effects. The user chooses the level of information that they wish to receive through the interactive interface, allowing for an individualized experience. Upon reaching the end of the tool, information on the tablet suggests that women ask their provider about HIV prevention methods they are interested in using, based on their preferences for method characteristics, and their questions to facilitate deliberation with the provider. The DST takes approximately 10 minutes to complete. A decision support tool was chosen as a key component of the study following its proven effectiveness in offering contraceptive options to patients. The HIV prevention DST was tested in Aim 1 of this study: participants were randomized to viewing the DST or not, prior to receiving usual care.

Additionally, the study team recognizes the importance of receiving health information from a trusted source, such as health care providers or health educators, when making important health decisions. Therefore, this study (Aim 2) will offer and assess the effects of a combined intervention of the DST following a clinic-wide training on shared decision making and trauma-informed care. Shared decision making is an effective strategy to offer information and services to patients as it allows the health care provider to share their clinical knowledge and expertise while partnering with the patient to elicit their experiential knowledge, needs and preferences. Through partnership between a patient and provider, the patient can make an informed decision about HIV prevention and other health needs that align with their values and desires and can result in greater adherence to the prevention or treatment options and satisfaction with care. The training will also include information about trauma-informed approaches to deliver health care in a person-centered and affirming manner. This training will highlight how many people, particularly those vulnerable to HIV due to intersecting oppressions, carry traumas that impact their exposure to health issues and the resources needed to mitigate these harms. It is critical that health care providers and health professionals are aware of intersecting forms of oppression that create trauma, including those that the medical profession create and perpetuate. A combined approach of shared decision making at the interpersonal level and trauma informed care at the clinic-level is an equity-oriented strategy to offering HIV prevention information to women in the Southeastern U.S. who are disproportionately impacted by HIV.

Approximately 366 individuals who self-identify as women presenting to one reproductive health clinic in Duval County, Florida, will be recruited to the study in Aim 2, with 183 enrolled in each of the two phases. As the decision support tool is primarily focused on cisgender women, participants who do not identify as cisgender will be included in the study, but their study data will be analyzed separately. In the first phase of Aim 2 of the study, participants will receive care as usual at a clinic site after the trainings have been held for staff. In the second phase of Aim 2, participants will receive care at this same clinic that has been exposed to the training and will also view the HIV prevention DST. These participants will be compared to those recruited in Aim 1 of this study, in which participants accessed care from the same clinic prior to clinic-wide trainings, and half of participants viewed the HIV prevention DST.

In addition to these interventions, a subset of 40 participants (20 per phase) will be asked to allow audio-recording of their counseling sessions with a provider. A subset of up to 40 additional participants (20 per phase), all of whom self-identify as women of color, will be invited to complete one-hour, semi-structured interviews after their clinic visit about their experiences of using the DST, HIV prevention counseling, and decision making about PrEP. Those who participated in Aim 1, are not excluded from participating in Aim 2 however, they will not be eligible to participate in an interview.

Hypotheses:

1. Women who receive care at a clinic following clinic-wide trainings on shared decision making and trauma informed care are more likely to initiate PrEP as compared to women who received care at the same clinic prior to training.
2. In a clinic that received clinic-wide trainings in shared decision making and trauma informed care, women who use the HIV prevention decision support tool are more likely to initiate PrEP as compared to women who did not use the tool.
3. Women who receive care at a clinic following clinic-wide training on shared decision making and trauma informed care and who also used the decision support tool are more likely to initiate PrEP as compared to women who receive care at the same clinic prior to training and did not use the tool.
4. Women who receive care at a clinic following clinic-wide trainings on shared decision making and trauma informed care and who also used the decision support tool are more likely to initiate PrEP as compared to those who receive care at the same clinic prior to training and used the DST.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as a woman (regardless of pregnancy status)
* Age 18 years - 45 years
* Not known to be living with HIV (based on self-report)
* English speaking
* Interested in participating in the study

Exclusion Criteria:

* Unable to consent
* Currently using PrEP
* Those who were assigned male at birth and self-identify as a man
* Unwilling to be contacted in 3 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Anyone who self identifies as a woman
Enrollment: 141 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
PrEP Prescriptions (As Measured by Chart Review) | 3 months post baseline visit
  The number of participants who received a PrEP prescription within 3 months of their baseline visit, obtained by chart extraction from the medical record. Outcome is dichotomous (Yes, received a PrEP prescription at initial visit/No, did not receive a PrEP prescription at initial visit).

SECONDARY OUTCOMES:
Number of Patients Reporting PrEP Use | 3 months post baseline visit
  Patients will be contacted at follow-up and asked if they took PrEP in the past 3 months regardless of where it was obtained. Outcome is dichotomous ("Yes", initiated PrEP within 3 months of initial visit/"No", did not initiate PrEP within 3 months of initial visit)
Change in Patient-Perceived HIV risk | Baseline, pre-intervention compared to immediately post baseline visit
  We will measure the change in HIV risk perception from pre- to post-visit at baseline. Response options include 4-point scale: 1 ("Not at all worried") to 4 ("Extremely worried").
Patient-Perceived HIV risk | Immediately post baseline visit
  Participants will be asked about how worried they are about getting HIV in the next 6 months. Response options include 4-point scale of 1 ("Not at all worried") to 4 ("Extremely worried").
PrEP Knowledge | Immediately post baseline visit
  Proportion of participants selecting the correct response to three questions. Response options for each item are different. Higher score represents higher knowledge.
Decisional Conflict - Total Score | Immediately post baseline visit
  16-item scale to measure decisional conflict. Response options range from 1-5 "strongly disagree" to "strongly agree". Mean score will be calculated, subtracted by 1, and multiplied by 25; scores range from 0 [no decisional conflict' to 100 [extremely high decisional conflict].Higher scores represent high decisional conflict.
Decisional Conflict - Uncertainty Subscore | Immediately post baseline visit
  Three items from the Decisional Conflict scale will measure uncertainty: "I am clear about the best choice for me", "I feel sure about what to choose", and "the decision is easy for me to make". Response options range from 1-5 "strongly disagree" to "strongly agree". Items will be reverse-coded. Mean scores will be calculated, subtracted by 1, and multiplied by 25; scores range from 0 [feels extremely certain about best choice] to 100 [feels extremely uncertain about decision]. Higher scores represent greater decision uncertainty.
Decisional Conflict - Informed Subscore | Immediately post baseline visit
  Three items from the Decisional Conflict scale will measure the informed subscale: "I know which options are available to me", "I know the benefits of each option", and "I know the risks and side effects of each option". Response options range from 1-5 "strongly disagree" to "strongly agree". Items will be reverse-coded. Mean scores will be calculated, subtracted by 1, and multiplied by 25; scores range from 0 [feels extremely informed] to 100 [feels extremely uninformed]. Higher scores represent a greater degree of feeling uninformed.
Decisional Conflict - Values Clarity Subscore | Immediately post baseline visit
  Three items from the Decisional Conflict scale will measure values clarity: "I am clear about which benefits matter the most to me", "I am clear about which risks and side effects matter most to me", and "I am clear about which is more important to me (the benefits or the risks and side effects." Response options range from 1-5 "strongly disagree" to "strongly agree". Items will be reverse-coded. Mean scores will be calculated, subtracted by 1, and multiplied by 25; scores range from 0 [feels extremely clear about personal values for benefits and risks/side effects] to 100 [feels extremely unclear about personal values].
Decisional Conflict - Support Subscore | Immediately post baseline visit
  Three items from the Decisional Conflict scale will measure support: "I have enough support from others to make a choice", "I am choosing without pressure from others", and "I have enough advice to make a choice". Response options range from 1-5 "strongly disagree" to "strongly agree". Items will be reverse-coded. Mean scores will be calculated, subtracted by 1, and multiplied by 25; scores range from 0 [feels extremely supported in decision making] to 100 [feels extremely unsupported in decision making].
Decisional Conflict - Effective Decision Subscore | Immediately post baseline visit
  Four items from the Decisional Conflict scale will measure effective decision: "I feel I have made an informed choice", "my decision shows what is important to me", "I expect to stick with my decision", and "I am satisfied with my decision". Response options range from 1-5 strongly disagree to strongly agree. Items will be reverse-coded. Mean scores will be calculated, subtracted by 1, and multiplied by 25; scores range from 0 [good decision] to 100 [bad decision].
Interpersonal Quality of HIV Prevention Care | Immediately post baseline visit
  Mean score of 4-item scale. Derived from the Person-Centered Contraceptive Care measure developed by the PI. Response options consist of 5-point Likert scale: 1 ("strongly disagree") to 5 ("strongly agree"). Scores will be dichotomized between 20 [excellent interpersonal quality of care] and less than 20 [poor interpersonal quality of care].
Interpersonal Quality of Health Services | Immediately post baseline visit
  Mean score of 4-item scale. Derived from the Person-Centered Contraceptive Counseling measure developed by the PI. Response options consist of 5-point Likert scale: 1 ("strongly disagree") to 5 ("strongly agree"). Scores will be dichotomized between 20 [excellent interpersonal quality of care] and less than 20 [poor interpersonal quality of care]. This measure will exclude HIV prevention care and focus on other services offered.
Intention to Use Any HIV Prevention Method | Immediately post baseline visit
  A one time, one item measure of plan to use HIV prevention method after the initial visit. Participants can select from "none", condoms, PrEP, PEP, treatment as prevention, regular HIV testing (inclusive of partner), "still thinking about my options", or other method.
Confidence in Decision to Use an HIV Prevention Method | Immediately post baseline visit
  A one-time, one-item measure of certainty of plan to use HIV prevention after the initial visit. Participants can select from four options: 1 ("completely unsure"), 2 ("mostly unsure"), 3 ("mostly sure, but not 100%"), or 4 ("100% sure").
Satisfaction with Information Received about HIV Prevention | Immediately post baseline visit
  Participants will be asked a one-time question regarding satisfaction with HIV prevention counseling. Response options include: 1 ("I was not given any information about HIV), 2 ("Very unsatisfied") 3 ("Somewhat unsatisfied), 4 ("Neither satisfied or unsatisfied"), 5 ("Somewhat satisfied") and 6 ("Very satisfied").
Perceived Quality of Information Received about HIV Prevention | Immediately post baseline visit
  Participants will also be asked four questions about the perceived quality of the HIV prevention information patients received during their health care visit: 1) getting the information they needed, 2) the ease of understanding the information, 3) the trustworthiness of the information, and 4), the usefulness of the information. These questions will be asked of those who reported talking about HIV/HIV prevention during their visit with the healthcare provider or health educator OR those who talked to the healthcare provider or health educator about your chances of getting HIV. Response options are 1 to 5 "strongly disagree" to "strongly agree". Higher values indicate greater perceived quality.
Perceived Quality of Health Information Received | Immediately post baseline visit
  Participants will also be asked four questions about the perceived quality of the health information patients received during their health care visit, excluding HIV prevention information: 1) getting the information they needed, 2) the ease of understanding the information, 3) the trustworthiness of the information, and 4), the usefulness of the information. These questions will be asked of those who reported talking about alcohol or drugs, intimate partner violence or abuse, pregnancy, contraception or birth control, STDs (not including HIV) or STD prevention, or other, during their visit with the healthcare provider or health educator. Response options are 1 to 5 "strongly disagree" to "strongly agree". Higher values indicate greater perceived quality.
Acceptability of HIV Prevention Methods | Immediately post baseline visit
  Participants are asked to rate their preference for a method (even if they never used it). Participants can select from condoms, PrEP, PEP, treatment as prevention or other method. The option, "never heard of it" is also included. Options for this scale range from 0 ("Terrible method for me") to 10 ("Great method for me").
Acceptability of the Decision Support Tool | Immediately post baseline visit
  Participants who used the DST in the second phase of the study are asked four questions about their experiences using the DST (e.g., degree to which they got all the information they needed, found the information to be easy to understand, trust the information, and found information useful). Response items vary from strongly disagree to strongly agree.
Perception of the Decision Support Tool | Immediately post baseline visit
  Participants who used the DST in the second phase of the study will be asked about the degree to which they liked/disliked the tool. Response options vary: "I did not like it at all", "I somewhat liked it", "I somewhat liked it", or "I really liked it".
Satisfaction with the Decision Support Tool | Immediately post baseline visit
  Participants who used the DST in the second phase of the study will be asked about the degree to which they are satisfied with the information in the tool. Response options vary from 1-5: "very unsatisfied" to "very satisfied".
Recommend the Decision Support Tool | Immediately post baseline visit
  Participants who used the DST in the second phase of the study will be asked about whether they would recommend the decision support tool to a friend. Response options are "yes", "no", and "unsure".
Willingness to Use the Decision Support Tool at Future Visits | Immediately post baseline visit
  Participants who used the DST in the second phase of the study will be asked about whether they would use the tool again if they returned to the clinic. Response options are "yes", "no", and "unsure"
HIV Prevention Method Use (any method - planned or new method) | 3 months post baseline visit
  A self-reported measure of HIV prevention method use, including those who reported discontinuing the initial HIV prevention method(s) that were reported post-clinic visit. This item will be measured by a response of "yes" to any of the following questions: since your [baseline] visit, have you used....for HIV prevention - abstinence, condoms, PEP, PrEP, regular HIV testing, treatment as prevention, regular sexually transmitted disease (STD) testing, or other method. The outcome will be dichotomized to those who responded affirmatively vs other responses ("no"/"unsure").
HIV Prevention Method Continuation | 3 months post baseline visit
  A self-reported measure of HIV prevention method continuation. This item will be measured by a response of "yes" to any of the following questions: are you still using - abstinence, condoms, PEP, PrEP, regular HIV testing, treatment as prevention, regular sexually transmitted disease (STD) testing, or other method. The outcome will be dichotomized to those who responded "yes" vs "no".

CONTACTS AND LOCATIONS:
Overall Officials: Christine Dehlendorf, MD, MAS, Principal Investigator — University of California, San Francisco; Akilah Pope, MD, Principal Investigator — Florida Department of Health, Duval County
Locations (1):
- Florida Department of Health, Duval County, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No